CLINICAL TRIAL: NCT03394014
Title: Ultrasound -Guided Sciatic Nerve Block in Below Knee Amputation Surgery: Subgluteal Versus Popliteal
Brief Title: Ultrasound-guided Sciatic Nerve Block in Below Knee Amputation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Maher Hussien, principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: FMASU R46/2017
Record Dates: First submitted 2017-12-24; First posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Sciatic Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- popliteal sciatic nerve block (Active Comparator): injecting 25 ml of bupivacaine 0.5 % (Sunnypivacaine, 20 ml vial contains Bupivacaine HCL Monohydrate 105.5 mg eq. to 100 mg Bupivacaine HCL, Sunny Pharmaceutical, Badr city- Cairo- Egypt) once circumferentially around the sciatic nerve at the popliteal fossa using ultrasound device (S-Nerve ultrasound system, Fujifilm Sonosite Inc., Bothell, WA)
  Interventions: Procedure: sciatic nerve block
- subgluteal sciatic nerve block (Active Comparator): injecting 25 ml of bupivacaine 0.5 % (Sunnypivacaine, 20 ml vial contains Bupivacaine HCL Monohydrate 105.5 mg eq. to 100 mg Bupivacaine HCL, Sunny Pharmaceutical, Badr city- Cairo- Egypt) circumferentially around the sciatic nerve at the subgluteal region using ultrasound device (S-Nerve ultrasound system, Fujifilm Sonosite Inc., Bothell, WA).
  Interventions: Procedure: sciatic nerve block

INTERVENTIONS:
Procedure: sciatic nerve block — blocking sciatic nerve either at the subgluteal area or the popliteal region for effective anesthesia and analgesia during below knee amputation
  Other Names: sciatic nerve block at the subgluteal and popliteal region

SUMMARY:
56 ASA physical status II and III patients, aged 45-75 year, undergoing elective below knee amputation were randomly assigned to receive either sciatic nerve block using a popliteal approach or a sub gluteal approach. Patients in both groups received same amount of LA and additional ultrasound guided femoral nerve block to ensure sensory block of the medial side of the leg. Success of the block was considered when the block is solid and doesn't require shifting to GA

DETAILED DESCRIPTION:
56 ASA physical status II and III patients, aged 45-75 year, undergoing elective below knee amputation were randomly assigned to receive either sciatic nerve block using a popliteal approach (group P, n 28) or a sub gluteal approach (group G, n 28). Patients in both groups received same amount of LA (25 ml of bupivacaine 0.5 %) and additional ultrasound guided femoral nerve block by 10 ml of bupivacaine 0.5% to ensure sensory block of the medial side of the leg. Time to complete sensory and motor block, time taken to perform the block, block-related complications, block duration, time for asking for rescue analgesia in the first 24 h were recorded and both patients and surgeons were asked about their level of satisfaction. Success of the block was considered when the block is solid and doesn't require shifting to GA

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status II and III patients
* aged 45-75 years,
* undergoing elective below knee amputation

Exclusion Criteria:

* patients who refused to participate in the study,
* those having allergy to local anaesthetics,
* or having contraindications to regional anaesthesia (having neurologic or neuromuscular disease, on anticoagulation therapy, or having skin infection at the site of needle insertion).

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
to compare between the two techniques as regards the success rate. | 24 hours
  Success was considered when the block provided solid analgesia with no need to shift to GA

SECONDARY OUTCOMES:
time taken to perform the block | 10-20 min
  time required to perform either block